CLINICAL TRIAL: NCT00000756
Title: Evaluation of the Safety and Tolerance of Immunotherapy With Autologous, Ex-Vivo Expanded, HIV-Specific Cytotoxic T-Cells in HIV-Infected Patients With CD4+ Counts Between 100-400/mm3
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: DATRI 006; 11736 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-03 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: T-Lymphocytes; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Immunotherapy, Adoptive; Transplantation, Autologous
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Lymphocyte Count

INTERVENTIONS:
Drug: Lymphocytes, Activated

SUMMARY:
To determine the safety, tolerance, and feasibility of adoptive immunotherapy with autologous cytotoxic T-lymphocytes (CTLs) in HIV-infected patients with CD4 counts between 100 and 400; to evaluate the immunologic, virologic, and clinical changes for up to 24 weeks following infusion of study therapy.

Freshly isolated peripheral blood lymphocytes from HIV-1-seropositive individuals frequently lyse autologous HIV-1-expressing cells or autologous cells infected with vaccinia vectors encoding HIV-1-specific proteins. Administration of these cytotoxic T lymphocytes (CTLs) may help prevent HIV disease progression.

DETAILED DESCRIPTION:
Freshly isolated peripheral blood lymphocytes from HIV-1-seropositive individuals frequently lyse autologous HIV-1-expressing cells or autologous cells infected with vaccinia vectors encoding HIV-1-specific proteins. Administration of these cytotoxic T lymphocytes (CTLs) may help prevent HIV disease progression.

AMENDED 03/28/94:

Patients are not accrued at the 25 billion CTL dose. Instead, a third cohort receives three infusions of 1 billion CTL 5-8 weeks apart.

AMENDED 02/14/94:

Patients infused with 1 or 5 billion CTL will be reinfused with 1 billion CTL 6-12 months later, and then followed for up to 12 weeks after the reinfusion.

ORIGINAL DESIGN:

Fifteen patients whose cells show an HIV-specific cytotoxic T lymphocyte (CTL) response are infused with autologous, ex-vivo expanded CTLs at a dose of 1, 5, or 25 billion cells (five patients per dose level). If one to three patients at a given dose develop acute toxicity, an additional three patients will be entered at that dose. If four patients at any given dose develop acute toxicity, the next lower dose will be designated as the MTD (if four patients develop acute toxicity in the first cohort, the study will be terminated). Patients are evaluated during infusion and at 1, 2, 4, 8, and 24 weeks.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Approved antiretroviral therapy and/or prophylactic PCP therapy, provided there was no change in such therapy in the 4 weeks prior to study entry.
* Other approved treatments for HIV-related diseases that are not known to affect cellular immune response.
* G-CSF.
* Erythropoietin.
* Supportive care for acute therapy-related toxicity.

Patients must have:

* HIV infection.
* CD4 count 100 - 400 cells/mm3.
* No current or previously documented AIDS-related opportunistic infection, malignancy, or encephalopathy other than mild Kaposi's sarcoma.
* FEV1 > 70 percent, DLCO > 50 percent predicted for height and age (initial infusion only).
* T cell lines with specific cytotoxicity against HIV-1.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Significant autoimmune disease.
* Non-AIDS-associated malignancy.
* Symptoms of cardiac disease.
* Dyspnea on significant exertion.
* Acute infiltrates on chest radiographs.

Patients with the following prior conditions are excluded:

* History of significant arrhythmia, infarction, or heart failure.
* History of a major psychiatric illness.

Prior Medication:

Excluded within 4 weeks prior to study entry:

* Systemic immunosuppressive therapy (i.e., steroids, cyclosporine, chemotherapy, or alpha-interferon).
* Therapy for acute infection, AIDS-related opportunistic infection, or malignancy.
* Experimental AIDS therapy.

Prior Treatment:

Excluded:

* Potentially immunosuppressive local therapy or radiation therapy for Kaposi's sarcoma within 4 weeks prior to study entry.

Current substance abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15
Dates: Study Completion 2002-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: J Lieberman, Study Chair; H Standiford, Study Chair; D Stein, Study Chair
Locations (1):
- New England Med Ctr / Tufts Univ, Boston, Massachusetts, United States

REFERENCES:
- [Background] Lieberman J, Skolnik PR, Parkerson GR 3rd, Fabry JA, Landry B, Bethel J, Kagan J. Safety of autologous, ex vivo-expanded human immunodeficiency virus (HIV)-specific cytotoxic T-lymphocyte infusion in HIV-infected patients. Blood. 1997 Sep 15;90(6):2196-206. PMID 9310470